CLINICAL TRIAL: NCT05866965
Title: Effect of Platelet-rich Fibrin on Soft Tissue, Periodontal Pocket Healing and Alveolar Bone Height After Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lam Cu Phong (Other)
Responsible Party: Sponsor-Investigator, Lam Cu Phong, Lecturer, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: lamphongrhm
Record Dates: First submitted 2023-04-27; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Platelet-rich Fibrin

STUDY DESIGN:
Intervention Model Description: split-mouth study, 1 side would be the study side and other side would be control side
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): standard third molar surgery following surgical protocol of Department of Oral Surgery, University of Medicine and Pharmacy
  Interventions: Other: standard third molar surgical removal
- PRF (Experimental): PRF was applied in third molar socket after removal following surgical protocol of Department of Oral Surgery, University of Medicine and Pharmacy
  Interventions: Other: PRF

INTERVENTIONS:
Other: PRF — centrifuge patient's blood to collect 1 block of yellowish condensed fibrin, which is platelet-rich fibrin
  Arms: PRF
Other: standard third molar surgical removal — standard third molar surgery following surgical protocol of Department of Oral Surgery, University of Medicine and Pharmacy
  Arms: control

SUMMARY:
A Randomized, controlled clinical trial and split-mouth design was performed to assess and compare the effect of platelet-rich fibrin (PRF) on soft tissue healing, periodontal pocket depth and alveolar bone height distal to second molar of the study and control groups after third molar surgical removal.

Sample include of participants who had indication of impacted lower third molars extraction on both sides with symmetrically orientation and same difficult index. All participants had same extraction protocol on both side at Department of Oral surgery, Faculty of Odonto-stomatology, University of Medicine and Pharmacy, Ho Chi Minh City.

Soft tissue healing, periodontal pocket depth and distal bone height were evaluation by an independent investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Good general health.
* Bilateral lower third molars equivalent in inclination and Pell and Gregory's impaction classification (classification II, III and B, C). The assessment of equivalence between two mandibular third molars was determined on the panoramic radiograph.
* The difference of third molar inclination on both sides not greater than 15 degrees.
* The patient consented to participate in the study after hearing clearly the explanation of purposes and requirements of the study.

Exclusion Criteria:

* Patients with any systemic disease contraindicated for surgery.
* Presence of acute inflammation or infection at third molar areas.
* Patients refused to participate in the study, did not comply with treatment or did not come to the follow-up examination as required.
* The difference in surgical time between the two groups was more than 10 minutes.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
periodontal pocket depth | 1rst postoperative month
  periodontal pocket depth at distal buccal and distal lingual side of second molar
periodontal pocket depth | 3rst postoperative month
  periodontal pocket depth at distal buccal and distal lingual side of second molar
periodontal pocket depth | 6rst postoperative month
  periodontal pocket depth at distal buccal and distal lingual side of second molar
distal bone resorption | 3rd postoperative month
  resorption of alveolar bone height distal to second molar
distal bone resorption | 6th postoperative month
  resorption of alveolar bone height distal to second molar

SECONDARY OUTCOMES:
soft tissue healing index | 3rd postoperative day
  soft tissue healing around third molar socket
soft tissue healing index | 7th postoperative day
  soft tissue healing around third molar socket

CONTACTS AND LOCATIONS:
Overall Officials: Phong Cu Lam, Master, Principal Investigator — University of Medicine and Pharmacy, Ho Chi Minh city
Locations (1):
- University of Medicine and Pharmacy, Ho Chi Minh City, Vietnam